CLINICAL TRIAL: NCT03631173
Title: Monitoring of patIents With Microdialysis Following Pancreaticoduodenectomy - a Randomized Controlled Trial. THE MINIMUM STUDY
Brief Title: Monitoring of patIents With Microdialysis Following Pancreaticoduodenectomy
Acronym: MINIMUM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Espen Lindholm, Senior researcher, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/1334
Record Dates: First submitted 2018-07-09; First posted 2018-08-15 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer; Pancreatic Neoplasms; Biliary Tract Cancer; Duodenal Cancer; Pancreatic Fistula
Keywords: Pancreaticoduodenectomy; Pancreatectomy; Anastomosis, Surgical
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms; Duodenal Neoplasms; Pancreatic Fistula | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: 2-armed, multicenter, randomized, open label, parallel-group controlled trial (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with microdialysis (Active Comparator): Intervention group - Patients will receive an intraperitoneal microdialysis catheter and will be monitored consecutively by microdialysis. The surgeon is familiar with the current microdialysis results at any time during the study period. The surgeon may intervene based on traditional symptoms and signs plus predetermined values of the microdialysis results.
  Interventions: Procedure: Surgical og radiological intervention, antibiotics
- Patient without microdialysis (No Intervention): The control group - The patients will not receive a microdialysis catheter. The patients are monitored according to current standards of care and the surgeon may intervene based only on traditional symptoms and signs.

INTERVENTIONS:
Procedure: Surgical og radiological intervention, antibiotics — Intervention might be a new drainage catheter, replacement of old drainage catheter, reoperation, somatostatin- and antibiotic administration.
  Arms: Patient with microdialysis

SUMMARY:
A pancreaticoduodenectomy is performed in patient with pancreatic cancer. The most common and serious complication is leakage between the intestine and the remnant pancreas after this procedure. It occurs in 20-30%. The result is often prolonged hospital and ICU stay, reoperations and deaths (3-5%). To detect a leakage early before the patient becomes seriously ill, thereby initiating treatment is therefore very important. By inserting a thin microdialysis catheter near the anastomosis between pancreas and intestine before closure of the abdominal wall, the investigators will analyze substances such as lactic acid, pyruvate, glycerol, etc. and if these substances may reveal anastomosis leakage at an early stage. Observational studies have shown that if a leakage occurs, glycerol concentration in the microdialysate will rise significant after few hours, and changes in lactic acid and pyruvate values will change as a sign of inflammation. The investigators want to conduct a randomized study comparing patients undergoing pancreaticoduodenectomy and using microdialysis in half of the included population.

DETAILED DESCRIPTION:
Anastomotic leakage after pancreaticoduodenectomy is a feared complication with substantial mortality and morbidity. Treatment of a postoperative pancreatic fistula can be difficult and management may range from a simple observation with or without percutaneous drainage, to the urgent need for reoperation and management of abdominal sepsis with organ failure and prolonged intensive care. To diagnose a pancreatic fistula may have a delay of several days. The risk of death and severe morbidity raises considerable from a biochemical pancreatic fistula compared to the most serious form, a grade C. Also, the cost of managing a patient with a fistula is 1.3-6 times more than a patient with no complications after PD.

Microdialysis is a promising tool in patients who undergoes pancreaticoduodenectomy for early detection of postoperative pancreatic fistula development. The technique may reveal an fistula before severe symptoms occur and before the complication gives the patient serious and life-threatening symptoms. Earlier intervention of the postoperative pancreatic fistula may lead to better prognosis, less reoperations and interventions and shorter stay at the ICU/hospital. By monitoring intraperitoneal metabolites (glycerol, lactate, pyruvate and glucose) close to the pancreaticojejunostomy, signs of a leakage may be discovered in few hours, thereby make it possible for early intervention and prevent developement of serious progression of morbidity. The investigators want to perform a randomized study where half of the patients will receive a microdialysis catheter implanted close to the pancreaticoduodenal anastomosis before closure of the abdomen. At certain timepoints postoperatively microdialysate will be analyzed for glycerol, lactate, pyruvate and glucose and the data will be used in the decisionmaking of diagnosing a pancreatic anastomosis leakage in addition to standard management. The other half of the patients will not receive a microdialysis catheter and the decisionmaking will only be based on standard management (ie. inflammation markers in blood samples, amylase in drainage fluid).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be scheduled for a pancreaticoduodenectomy
* Subject must be ≥ 18 years
* Able to give written signed informed consent
* Investigator's assessment that the patient is able to understand, comply and follow the instructions needed to successfully participate in this trial

Exclusion Criteria:

* Allergic to Voluven® (Fresenius Kabi AS, Halden, Norway) and contrast given during CT scan
* Another study interfering with current study
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Total hospital stay | 30 days after surgery - postoperative day 30
  Number of days from end of surgery to hospital discharge (at any hospital)

SECONDARY OUTCOMES:
Length of stay at the primary hospital | 30 days after surgery - postoperative day 30
  Length of stay at the primary hospital and ICU. Number of days from initial operation to primary hospital discharge.
Concentration of Lactate (mM), Pyruvate (microM), Glycerol (microM), Glucose (mM) in microdialysate | 30 days after surgery - postoperative day 30
  Concentration of Lactate, Pyruvate, Glycerol, Glucose in microdialysate in relation to patients with or without anastomosis leakage
Concentration of inflammatory markers in microdialysate | 30 days after surgery - postoperative day 30
  Concentration of inflammatory markers in microdialysate in relation to patients with or without anastomosis leakage
Concentration of inflammatory markers in serum | 30 days after surgery - postoperative day 30
  Concentration of inflammatory markers in serum in relation to patients with or without anastomosis leakage
Patient-reported quality of life questionnaire - total score assessed by the Abdominal surgery Impact scale by summing subscores | From inclusion to 90-days after surgery
  Total score - Abdominal surgery Impact scale. The summative scores for the scale range from 18 to 126, with higher scores indicating better quality of life
Patient-reported quality of life questionnaire - subgroup score Physical limitations assessed by the Abdominal surgery Impact scale | From inclusion to 90-days after surgery
  Subgroup score Physical limitations - Abdominal surgery Impact scale. The summative scores for the scale range from 3 to 18, with higher scores indicating better physical ability
Patient-reported quality of life questionnaire - subgroup score Functional impairment assessed by the Abdominal surgery Impact scale | From inclusion to 90-days after surgery
  Subgroup score Functional impairment - Abdominal surgery Impact scale. The summative scores for the scale range from 3 to 18, with higher scores indicating better functional ability
Patient-reported quality of life questionnaire - subgroup score Pain assessed by the Abdominal surgery Impact scale | From inclusion to 90-days after surgery
  Subgroup score Pain - Abdominal surgery Impact scale. The summative scores for the scale range from 3 to 18, with higher scores indicating more pain
Patient-reported quality of life questionnaire - subgroup score Visceral Function assessed by the Abdominal surgery Impact scale | From inclusion to 90-days after surgery
  Subgroup score Visceral Function - Abdominal surgery Impact scale. The summative scores for the scale range from 3 to 18, with higher scores indicating more Visceral dysfunction
Patient-reported quality of life questionnaire - subgroup score Sleep assessed by the Abdominal surgery Impact scale | From inclusion to 90-days after surgery
  Subgroup score Sleep - Abdominal surgery Impact scale. The summative scores for the scale range from 3 to 18, with higher scores indicating more sleep dysfunction
Patient-reported quality of life questionnaire - subgroup score Psychological function assessed by the Abdominal surgery Impact scale | From inclusion to 90-days after surgery
  Subgroup score Psychological function - Abdominal surgery Impact scale. The summative scores for the scale range from 3 to 18, with higher scores indicating more psychological dysfunction
Patient-reported pain questionnaire - total score assessed by the McGill Pain Questionnaire-2 (SF-MPQ-2) | From inclusion to 90-days after surgery
  Total score - McGill Pain Questionnaire-2 (SF-MPQ-2). Subgroup score Psychological function - Abdominal surgery Impact scale. The summative scores ranging from 0 to 45, with higher score indicating more pain
Expenses (Euros) per patient used during total hospital stay | 30 days after surgery - postoperative day 30
  Number of Euros used in patient undergoing pancreaticoduodenectomy With or without microdialysis catheter
Daily assessement of microdialysis catheter malfunction during admission at hospital, at an average of 10 days after surgery | From surgery end to discharge from primary hospital, at an average of 10 days after surgery
  Number of catheter which are not functioning
Risk factors of postoperative pancreatic fistula at discharge from hospital, at an average 10 days after surgery | From surgery end to discharge from primary hospital at hospital, at an average of 10 days after surgery
  Numbers of risk factors of postoperative pancreatic fistula in relation to patients with or without anastomosis leakage
Risk factors of postoperative pancreatic fistula at 30 days after surgery | From surgery end to 30 days after surgery
  Numbers of risk factors of postoperative pancreatic fistula in relation to patients with or without anastomosis leakage
Risk factors of postoperative pancreatic fistula at 90 days after surgery | From surgery end to 90 days after surgery
  Numbers of risk factors of postoperative pancreatic fistula in relation to patients with or without anastomosis leakage

OTHER OUTCOMES:
Time before postoperative fistula is diagnosed (hours) | End of surgery to 30 days postoperative
  Hours from end of surgery to diagnosis of postoperative pancreatic fistula
Total quantity (μg/mg) of vasoactive medications at discharge at an average of 10 days after surgery | From surgery end to discharge from primary hospital at an average of 10 days after surgery
  Amount of vasoactive medication during surgery and postoperatively until discharge from the hospital where the surgery was performed.
Number of patients with Pancreatic Fistula | 30 days after surgery - postoperative day 30
  Number of patients with Pancreatic Fistula
Number of patients with Biliary Fistula | 30 days after surgery - postoperative day 30
  Number of patients with Biliary Fistula
Number of patients with gastroenteric Fistula | 30 days after surgery - postoperative day 30
  Number of patients with gastroenteric Fistula
Daily measurements during hospital admission of pancreatic amylase (U/L) and bilirubin (µmol/L ) concentrations in drainage fluid and in serum, at an average og 10 days after surgery | From surgery end to discharge from primary hospital at an average of 10 days after surgery
  Pancreatic amylase and bilirubin concentrations in drainage fluid and in serum
Postoperative complications | From inclusion to 90-days after surgery
  Number of patients with postoperative complications during total hospital stay
Fluid Balance (ml) during hospital admission at an average of 10 days after surgery | From anesthesia start to discharge from primary hospital at an average of 10 days after surgery
  Diuresis and amount of fluid given i.v. during surgery and postoperatively until discharge from the primary hospital
Number of patients discharged to home/self care at an average of 10 days after surgery | At discharge at an average of 10 days after surgery
  Patient's discharge disposition - number of patients Discharged to home/self care
Number of patients discharged to home but with home health service at an average of 10 days | At discharge at an average of 10 days after surgery
  Patient's discharge disposition - number of patients Discharged to home but with home health service
Number of patients discharged/transferred to nursing home at an average of 10 days | At discharge at an average of 10 days after surgery
  Patient's discharge disposition - number of patients Discharged/transferred to nursing home
Number of patients discharged/transferred to an inpatient rehabilitation facility at an average of 10 days | At discharge at an average of 10 days after surgery
  Discharged to an inpatient rehabilitation facility
Number of patients expired at an average of 10 days | At discharge at an average of 10 days after surgery
  Patient's discharge disposition - expired

CONTACTS AND LOCATIONS:
Overall Officials: Espen Lindholm, ph.d, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
No plan for individual participant data (IPD).

REFERENCES:
- [Derived] Lindholm E, Ekiz N, Tonnessen TI. Monitoring of patients with microdialysis following pancreaticoduodenectomy-the MINIMUM study: study protocol for a randomized controlled trial. Trials. 2021 May 7;22(1):329. doi: 10.1186/s13063-021-05221-9. PMID 33962656